CLINICAL TRIAL: NCT01424059
Title: Planned Induction of Women With Fear of Labor and Evaluation of the Experience of Delivery
Brief Title: Induction of Women With Fear of Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Maria Jonsson, M.D., Ph.D. Consultant, Uppsala University Hospital
Other Study IDs: UAS-11
Record Dates: First submitted 2011-08-05; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Fear
Keywords: fear; labor; induction; amniotomy; WEDQ-B; parous; cesarean section
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fear of labor: Parous women with fear of labor
  Interventions: Other: WEDQ-B (questionnaire)

INTERVENTIONS:
Other: WEDQ-B (questionnaire) — Questionnaires are answered after delivery; within 48 hours and after five weeks

SUMMARY:
The purpose of this study is to evaluate the experience of labor in parous women induced because of fear of labor and, to compare the experience of parous women induced without fear of labor. A comparison with the experience of women delivered with elective cesarean section because of fear of labor is done.

In the induced labors, the induction method is amniotomy. Between groups the experience of delivery is evaluated with a questionnaire: Wijma Delivery Expectancy Questionnaire(WEDQ-B).

Groups are also compared with regard to time from induction to delivery and rate of operative delivery.

Hypotheses:

* there is no difference in experience of delivery
* there is no difference in time to delivery or rate of operative deliveries

ELIGIBILITY:
Inclusion Criteria:

* parous
* induction or cesarean section
* amniotomy

Exclusion Criteria:

* non proficiency in the Swedish language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parous women with cercvical status allowing amniotomy as method for induction. Parous women planned for cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
experience of delivery | Within 48 hours after delivery
  Experience of labor is evaluated with a questionnaire (WEDQ-B) within 48 hours

SECONDARY OUTCOMES:
Operative delivery | within 48 hours
  within 48 hours from inclusion in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Akademiska hospital, Uppsala, Sweden